CLINICAL TRIAL: NCT04647149
Title: Effects of Early and Delayed Time-Restricted Eating on Body Weight and Metabolic Parameters in Adults With Overweight and Obesity
Brief Title: Effects of Early and Delayed Time-restricted Eating in Adults With Overweight and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Alvaro Reischak-Oliveira, Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRE_UFRGS#
Record Dates: First submitted 2020-11-14; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Time Restricted Feeding; Intermittent Fasting; Obesity; Overweight and Obesity
MeSH Terms: conditions — Intermittent Fasting; Obesity; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early Time-Restricted Eating (Experimental): 8-hour eating window between 08:00 and 16:00
  Interventions: Behavioral: Dietary Approach
- Delayed Time-Restricted Eating (Experimental): 8-hour eating window between 12:00 and 20:00
  Interventions: Behavioral: Dietary Approach
- Control (Experimental): 12-hour eating window between 08:00 and 20:00
  Interventions: Behavioral: Dietary Approach

INTERVENTIONS:
Behavioral: Dietary Approach — Dietary approaches with energy restriction performed at different times of the day.

SUMMARY:
Time-restricted eating (TRE) is a dietary approach that aims to increase fasting time and decrease the eating window. Promising TRE effects on weight loss and some cardiometabolic risk factors have been reported. However, there is a lack of randomized clinical trials that directly investigate the effect of TRE at different times of the day (early vs. delayed) in individuals with overweight and obesity. The present study investigates the effects of 8 weeks of TRE performed at different moments of the day on body composition and cardiometabolic parameters in adults with overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Male and female;
* Body mass index (BMI) between 25 and 34.9 kg/m²;
* Age between 20 and 40 years;
* Not engaged in any structured exercise program;
* Weight stable for ~3 months prior to the beginning of the study;
* Able to give written informed consent.

Exclusion Criteria:

* Current smoker;
* Cardiometabolic diseases (dyslipidemia, diabetes, hypertension, etc);
* Current treatment with medication or supplements which significantly affect the main studied variables;
* Night-shift workers;
* Night eating syndrome;
* Irregular sleep patterns;
* For women: pregnancy, planned pregnancy (within the study period), lactating or menopause;
* Habitual fasting window >16 hours;
* Concomitant participation in other studies.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Insulin resistance (indices) | Change from baseline. Measured at baseline and after 8 weeks.
  Including but not limited to Homeostatic Model Assessment for Insulin Resistance (HOMA-IR).
Fasting insulin levels (µIU/mL) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by enzyme-Linked Immunosorbent Assay
Fasting glucose levels (mg/dL) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by colorimetric method
Insulin Sensitivity (indices) | Change from baseline. Measured at baseline and after 8 weeks.
  Including but not limited to the Matsuda index
Glucose tolerance | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by oral glucose tolerance test (OGTT; 0,30,60,90, and 120 min)
Fasting lipid profile levels (mg/dL) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by colorimetric method

SECONDARY OUTCOMES:
β cell function (indices) | Change from baseline. Measured at baseline and after 8 weeks.
  Including but not limited to HOMA-BETA
Fat Mass (kg) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by Dual-energy X-ray Absorptiometry under fasting condition.
Fat Percentage (%) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by Dual-energy X-ray Absorptiometry under fasting condition.
Fat Free Mass (kg) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by Dual-energy X-ray Absorptiometry under fasting condition.
Body Weight (kg) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by Dual-energy X-ray Absorptiometry under fasting condition.
Body Weight (kg) | Change from baseline. Measured at baseline and after 4, and 8 weeks.
  Measured on a digital scale.
Bone Mineral Content (kg) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by Dual-energy X-ray Absorptiometry under fasting condition.
Body Mass Index (kg/m^2) | Change from baseline. Measured at baseline and after 8 weeks.
  Calculated from weight in kilograms divided by height in meters squared.
Fasting ketones (β-hydroxybutyrate) levels (mmol/L) | Change from baseline. Measured at baseline and after 8 weeks.
Resting metabolic rate (Kcal/day) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by indirect calorimetry under resting and fasting conditions.
Substrate Oxidation (respiratory exchange ratio) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by indirect calorimetry under resting and fasting conditions.
Peak oxygen consumption (mL/min and mL/kg/min) | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by an open-circuit spirometry system
Quality of sleep | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by Pittsburgh Sleep Quality Index Questionnaire. Higher scores indicate worse sleep quality.
Risk of binge eating | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by binge eating scale. Higher scores indicate greater risk of binge eating.
Subjective appetite parameters (hunger, fullness, prospective food consumption, and desire to eat). | Change from baseline. Measured at baseline and after 8 weeks.
  Measured by visual analog scale.The scale range is 0-100 mm and each end represent the extremes.

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Reischak-Oliveira, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil